CLINICAL TRIAL: NCT02882113
Title: Influence of CYP3A5 Polymorphism on Liver Function Abnormality and the Trough Level Change After Conversion From Tacrolimus (Bid) to Advagraf® (qd) in Stable Liver Transplant Recipients
Brief Title: Influence of CYP3A5 Polymorphism on Liver Function Abnormality and the Trough Level Change After Conversion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKR-ADVLT-2014-02
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-06

CONDITIONS: Liver Dysfunction
MeSH Terms: conditions — Liver Diseases | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expressor (Experimental): CYP3A5 expressor; containing CYP3A5*1 wild-type allele(*1/*1 type & *1/*3 type) intervention: Advagraf conversion
  Interventions: Drug: Advagraf
- Non-expressor (Active Comparator): CYP3A5 non-expressor: without CYP3A5*1 allele( *3/*3 type) intervention: Advagraf conversion
  Interventions: Drug: Advagraf

INTERVENTIONS:
Drug: Advagraf — same dose as Tacrolimus bid der day in 24 weeks
  Other Names: Tacrolimus

SUMMARY:
This study is a multicenter, single-arm, open-label, 24 weeks, and investigator-initiated clinical trial to assess the influence of CYP3A5 polymorphism on liver function abnormality and the trough level change after conversion to Advagraf® in liver transplant recipients.

DETAILED DESCRIPTION:
All subjects who are liver transplant recipients taking Tacrolimus bid and adaptable to be registered for the study will be classified by expressive or non-expressive CYP3A5 polymorphism genotype and Advagraf® will be administered same dose as Tacrolimus bid der day in 24 weeks.

All subjects should check whether being registered in the hospital based on CYP3A5 polymorphism genotype during screening visit. Registered subjects will visit seven times to the hospital during the study which includes screening visit and adverse reaction, acute rejection, and trough level will be tested during this period. Subjects who are additionally agreed for PK study will be hospitalized with the state of Tacrolimus bid therapy one day ago before taking IP. On the first day of hospitalization, his/her blood will be collected. At week 1 (plus seven days) after conversion to Advagraf®, his/her blood will be collected for PK analysis.

ELIGIBILITY:
Inclusion Criteria:

* 19 years old and above.
* Patients who previously have received a liver transplant over the last six months and within last three years.
* Patients who are on Tacrolimus immunosuppressive therapy twice a day for at least two weeks.
* During Tacrolimus immunosuppressive therapy twice a day for at least two weeks, patients who have following conditions.

  * Patients who have normal liver function and renal function.
  * Patients who have been monitored without complication such as acute rejection.
* Patients willing to sign his/her consent.

Exclusion Criteria:

* Patients who have Tacrolimus trough level resulted as 2 ng/mg at the baseline.
* Patients who are on steroid therapy due to positive result of acute rejection test before the baseline.
* Patients who have received a transplant besides liver.
* Patients who are allergic to IP or macrolide compounds.
* Patients who are on cyclosporine, bosentan, or potassium sparing diuretic.
* Patients with genetic diseases such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
* Pregnant or lactating women.
* Patients not willing to adhere to study procedures/treatments.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
liver function abnormality rate | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-Woong Lee, Dr., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim JM, Ryu JH, Lee KW, Hong SK, Yang K, Choi GS, Kim YA, Lee JY, Yi NJ, Kwon CHD, Chu CW, Suh KS, Joh JW. Effect of CYP3A5 on the Once-Daily Tacrolimus Conversion in Stable Liver Transplant Patients. J Clin Med. 2020 Sep 8;9(9):2897. doi: 10.3390/jcm9092897. PMID 32911703